CLINICAL TRIAL: NCT05113966
Title: A Phase 2, Single-Arm, Open-Label Study of Trilaciclib Administered Prior to Sacituzumab Govitecan-hziy in Patients With Unresectable Locally Advanced or Metastatic Triple-Negative Breast Cancer Who Received at Least Two Prior Treatments, at Least One in the Metastatic Setting
Brief Title: Trilaciclib in Patients Receiving Sacituzumab Govitecan-hziy for Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor decided to close enrollment to the study on Feb 14, 2023, in order to reallocate resources to other ongoing trilaciclib clinical trials.
Sponsor: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G1T28-213
Record Dates: First submitted 2021-10-18; First posted 2021-11-09 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-11

CONDITIONS: Triple Negative Breast Cancer
Keywords: TNBC; Trodelvy; Myelosuppression
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — trilaciclib; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Trilaciclib + Sacituzumab Govitecan-hziy (Experimental): Participants received trilaciclib + sacituzumab govitecan-hziy on days 1 & 8 of a 21 day cycle. Trilaciclib is administered first, followed by sacituzumab govitecan-hziy. Administer diluted trilaciclib solution as a 30-minute IV infusion to be completed within 4 hours prior to the start of sacituzumab govitecan-hziy.
  Interventions: Drug: Trilaciclib; Drug: Sacituzumab Govitecan-hziy

INTERVENTIONS:
Drug: Trilaciclib — Single-use, sterile powder to be reconstituted and further diluted with 250 milliliters (mL) of normal saline (sodium chloride solution 0.9%) or dextrose 5% in water (D5W)
  Other Names: G1T28; CDK 4/6 inhibitor
Drug: Sacituzumab Govitecan-hziy — 10 milligram per kilogram (mg/kg) reconstituted to a concentration of 1.1 mg/mL to 3.4 mg/mL in normal saline
  Other Names: Trodelvy; IMMU-132

SUMMARY:
This was a Phase 2, multicenter, open-label, single-arm study evaluating the safety and efficacy of trilaciclib administered prior to sacituzumab govitecan-hziy in participants with unresectable, locally advanced or metastatic triple-negative breast cancer (TNBC) who received at least 2 prior treatments, at least 1 in the metastatic setting.

DETAILED DESCRIPTION:
The study included 3 study phases: Screening Phase, Treatment Phase, and Survival Follow-up Phase. The Treatment Phase began on the day of the first dose of study treatment and was completed at the Safety Follow-up Visit. Trilaciclib and sacituzumab govitecan-hziy were administered intravenously (IV) in 21-day cycles. Study drug administration continued until progressive disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or clinical progression as determined by the Investigator, unacceptable toxicity, withdrawal of consent, Investigator decision, or the end of the study, whichever occurred first. The first Survival Follow-up assessment occurred approximately 3 months after the Safety Follow-Up Visit and continued every 3 months until the end of the study (or death).

ELIGIBILITY:
Inclusion Criteria:

1. Adult ( ≥18 years of age), female or male participant with measurable (per RECIST v1.1), unresectable locally advanced or metastatic TNBC
2. Documentation of histologically or cytologically confirmed ER-negative, PR-negative, and HER2-negative tumor per the American Society of Clinical Oncology (ASCO) and the College of American Pathologists (ASCO/CAP) criteria.
3. Measurable disease as defined by RECIST v1.1.
4. Considered to be eligible to receive sacituzumab govitecan-hziy treatment, in the Investigator's judgment.
5. Participants must have received 2 or more prior lines of systemic therapy, at least one of them in the metastatic setting.
6. Radiation therapy for metastatic disease is permitted as long as the participant has at least 1 measurable lesion that has not been irradiated. Participants should be sufficiently recovered from the effects of radiation as determined by the Investigator but must have completed radiotherapy at least 2 weeks prior to enrollment.
7. ECOG performance status of 0 or 1.
8. Adequate organ function as demonstrated by the following laboratory values:

   * Hemoglobin ≥9.0 g/dL
   * Absolute neutrophil count (ANC) ≥1.5 × 10^9/L;
   * Platelet count ≥100 × 10^9/L;
   * Estimated glomerular filtration rate ≥30 mL/minute/1.73 m^2;
   * Total bilirubin ≤1.5 × upper limit of normal (ULN);
   * ALT and AST ≤3 × ULN in the absence of liver metastasis or ≤5 × ULN in the presence of liver metastasis.
9. Resolution of nonhematologic toxicities from prior systemic therapy, radiation therapy, or surgical procedures to Common Terminology Criteria for Adverse Events (CTCAE) ≤ Grade 1 (except alopecia or peripheral neuropathy that may be Grade 2 or less).
10. Predicted life expectancy of ≥3 months.
11. Contraceptive use by men or women should be consistent with local guidelines regarding the methods of contraception for those participating in clinical studies.
12. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol.

Exclusion Criteria:

1. Prior treatment with trilaciclib, sacituzumab govitecan-hziy, irinotecan, Trop-2 antibody drug conjugate, or any therapy with a topoisomerase-1 payload.
2. Participants with known brain metastasis at enrollment.
3. Participants with known Gilbert's disease or known homozygous for the UGT1A1*28 allele.
4. Participants with bone-only disease.
5. Malignancies other than TNBC within 3 years prior to enrollment. Participants with malignancies of a negligible risk of metastasis or death (e.g., risk of metastasis or death <5% at 5 years as determined by the Investigator) are eligible provided they meet all of the following criteria:

   1. Malignancy treated with expected curative intent (e.g., adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent);
   2. No evidence of recurrence or metastasis by follow-up imaging and any disease-specific tumor markers.
6. History of clinically significant gastrointestinal bleeding, intestinal obstruction, or gastrointestinal perforation within 6 months of enrollment.
7. Receipt of any investigational medication within 4 weeks, or at least 5 half-lives, whichever is greater, prior to the first dose of study treatment.
8. Receipt of any cytotoxic chemotherapy within 2 weeks or antibody treatment for cancer within 3 weeks prior to the first dose of study treatment.
9. Receipt of any high dose systemic corticosteroids within 2 weeks prior to the first dose of study treatment.

   1. Low dose corticosteroids (≤20 mg prednisone or equivalent daily) are permitted if the dose is stable for 4 weeks, or if medically indicated as part of their pre-medications for infusions.
   2. Topical steroids and corticosteroid inhalers are allowed.
10. Current use of immunosuppressive medication, except for the following:

    1. Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
    2. Systemic corticosteroids at physiological doses ≤10 mg/day of prednisone or equivalent;
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
11. Use of oral or IV antibiotics within 2 weeks prior to enrollment.
12. QT corrected interval using Fridericia's formula (QTcF) >480 msec at screening (confirmed on repeat). For participants with ventricular pacemakers, QTcF >500 msec.
13. Uncontrolled ischemic heart disease or uncontrolled symptomatic congestive heart failure (Class III or IV as defined by the New York Heart Association functional classification system).
14. History of stroke or cerebrovascular accident within 6 months prior to first dose of study treatment.
15. Known serious active infection such as, but not limited to, human immunodeficiency virus (HIV) (e.g., viral load indicative of HIV, HIV 1/2 antibodies), Hepatitis B (e.g., Hepatitis B surface antigen reactive or Hepatitis B DNA detected), Hepatitis C (e.g., Hepatitis C ribonucleic acid [quantitative] is detected) or tuberculosis.
16. Severe infection within 4 weeks prior to enrollment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
17. Other uncontrolled serious chronic disease or psychiatric condition that in the Investigator's opinion could affect participant safety, compliance, or follow-up in the protocol.
18. Known hypersensitivity or allergy to irinotecan, SN-38, trilaciclib, or sacituzumab govitecan-hziy or any excipients of the aforementioned medications
19. Prior hematopoietic stem cell or bone marrow transplantation.
20. Pregnant or lactating women
21. Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study.
22. Received a live, attenuated vaccine within 4 weeks prior to the first dose of study treatment or anticipation that such a vaccine will be required during the study treatment period:

    a. Influenza vaccination should be given during influenza season only (approximately October through May in the Northern Hemisphere).
23. Legal incapacity or limited legal capacity.
24. Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or participants who are employees of G1 Therapeutics, Inc. directly involved in the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2024-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Conduct, Study Director — G1 Therapeutics, Inc.
Locations (22):
- United States (22):
  - Ironwood Physicians, Chandler, Arizona
  - Comprehensive Blood & Cancer Center, Bakersfield, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - UCLA Hematology/Oncology Parkside, Santa Monica, California
  - PIH Health, Whittier, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Memorial Healthcare System, Hollywood, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Duly Health and Care, Joliet, Illinois
  - New England Cancer Specialists, Scarborough, Maine
  - Minnesota Oncology Hematology, P.A., Woodbury, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Northwest Cancer Specialists, PC, Tigard, Oregon
  - Texas Oncology - Austin Central, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Longview Cancer Center, Longview, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc, Roanoke, Virginia
  - Multicare Health System, Auburn, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from Q4 2021 until Q2 2024 in 20 different centers.
Pre-assignment Details: The study included 3 study phases: Screening Phase, Treatment Phase, and Survival Follow-up Phase. The Treatment Phase began on the day of the first study treatment dose and was completed at the Safety Follow-up Visit. The first Survival Follow-up assessment occurred approximately 3 months after the Safety Follow-Up Visit.
Groups:
- Trilaciclib + Sacituzumab Govitecan-hziy: Participants received trilaciclib + sacituzumab govitecan-hziy on Days 1 and 8 of a 21-day cycle. Trilaciclib was administered first, followed by sacituzumab govitecan-hziy. Administer diluted trilaciclib solution as a 30-minute IV infusion completed within 4 hours prior to the start of sacituzumab govitecan-hziy.
  Trilaciclib: Single-use, sterile powder reconstituted and further diluted with 250 mL of normal saline (sodium chloride solution 0.9%) or D5W Sacituzumab Govitecan-hziy: 10 mg/kg reconstituted to a concentration of 1.1 mg/mL to 3.4 mg/mL in normal saline
Period: Overall Study
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Started | 30
Completed | 0
Not Completed | 30
Not completed — Death | 21
Not completed — Study Terminated by Sponsor | 9

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): included all enrolled participantswho were administered at least 1 dose of study drug.
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (11.09)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex at Birth: Female | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival was defined as the time (months) from the date of the first dose of the study drug to the date of documented radiographic disease progression per RECIST v1.1 or death due to any cause, whichever comes first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to approximately 23 months
Population: FAS: included all enrolled participants who were administered at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 30
months | 4.1 [2.2 to 7.3]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with the best overall response of confirmed complete response or confirmed partial response per RECIST v1.1 Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to approximately 24 months
Population: The Response Evaluable (RE) population included all participants who were in the FAS and who had measurable (target) tumor lesion(s) at the baseline tumor assessment and either (i) had at least 1 post-baseline tumor assessment, or (ii) do not have post-dose tumor assessment but had clinical progression as noted by the Investigator, or (iii) died due to disease progression prior to their first post-baseline tumor scan.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 30
percentage of participants | 23.3 [9.9 to 42.3]

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants with the best overall response of confirmed complete response, confirmed partial response, or stable disease lasting 24 weeks or longer since the first date of study drug administration per RECIST v1.1
Time Frame: Up to approximately 24 months
Population: RE: population included all participants who were in the FAS and who had measurable (target) tumor lesion(s) at the baseline tumor assessment and either (i) had at least 1 post-baseline tumor assessment, or (ii) did not have post-dose tumor assessment but had clinical progression as noted by the Investigator, or (iii) died due to disease progression prior to their first post-baseline tumor scan.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 30
percentage of participants | 46.7 [28.3 to 65.7]

4. Secondary Outcome: Duration of Objective Response (DOR)
Description: DOR was the time between the first objective response of CR or PR (confirmed) and the first date that progressive disease was documented or death, whichever comes first. DOR was only analyzed for the patients who had achieved objective responses.
Time Frame: Up to approximately 24 months
Population: The Response Evaluable (RE) population included all participants who were in the FAS and who had measurable (target) tumor lesion(s) at the baseline tumor assessment and either (i) had at least 1 post-baseline tumor assessment, or (ii) did not have post-dose tumor assessment but had clinical progression as noted by the Investigator, or (iii) died due to disease progression prior to their first post-baseline tumor scan. DOR was only analyzed for the participants who had achieved OR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 7
months | 8.8 [4.0 to NA] — Not evaluable due to the low number of responders.

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (months) from the date of the first dose of the study drug to the date of death for participants who died in the study due to any cause or the time to the last contact date known to be alive for those participants who survived as of the data cutoff date for the planned OS analysis (censored cases).
Time Frame: Up to approximately 24 months
Population: FAS: included all enrolled participants who were administered at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 30
months | 15.9 [9.9 to 20.9]

6. Secondary Outcome: Number of Participants With Occurrence of Severe Neutropenia (SN)
Description: Occurrences of SN in Cycles 1 and 2 and the overall study are reported.
Time Frame: Up to approximately 24 months
Population: FAS: included all enrolled participants who were administered at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 30
Participants
  Participants with At Least 1 Event During Cycles 1-2: No | 29
  Participants with At Least 1 Event During Cycles 1-2: Yes | 1
  Participants with At Least 1 Event During Overall Study: No | 29
  Participants with At Least 1 Event During Overall Study: Yes | 1

7. Secondary Outcome: Participants With At Least One Occurrence of Febrile Neutropenia (FN)
Description: FN was defined as a complication of cancer treatment. It is the development of a fever, alongside other signs of infection such as feeling unwell, shivers, and shakes in a participant with neutropenia.
Time Frame: Up to approximately 24 months
Population: FAS: included all enrolled participants who were administered at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 30
Participants
  No | 29
  Yes | 1

8. Secondary Outcome: Occurrence of Granulocyte Colony-stimulating Factor (G-CSF) Administration
Description: The number of cycles with G-CSF administrations for a participant was the total number of cycles where the participant received at least one dose of G-CSF, for participants who did not have any G-CSF use and those who were enrolled but did not receive any study treatment, a value of 0 was assigned.
Time Frame: Up to approximately 24 months
Population: FAS: included all enrolled participants who were administered at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 30
Participants
  Participants with At Least One Event - No | 23
  Participants with At Least One Event - Yes | 7

9. Secondary Outcome: Occurrence of Grade 3 or 4 Decreased Hemoglobin (Hgb)
Description: The occurrence of Grade 3 or 4 decreased hemoglobin (Hgb) for a participant was defined as having at least one Hgb value that was < 8.0 gram per deciliter (g/dL) among all scheduled or unscheduled assessments. It was a binary random variable (Yes or No).
Time Frame: Up to approximately 24 months
Population: FAS: included all enrolled participants who were administered at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 30
Participants
  No | 30
  Yes | 0

10. Secondary Outcome: Number of RBC Transfusions
Description: Based on the NCCN Clinical Practice Guidelines in Oncology for Hematopoietic Growth Factors Version 2.2020 and the AABB Clinical Practice Guidelines, the following RBC transfusion thresholds were recommended; however, the participant's clinical situation should always be the primary guiding factor when deciding to transfuse.
  * Transfusion is not indicated until the hemoglobin level is ≤7 g/dL for hospitalized adult hemodynamically stable participants .
  * An RBC transfusion threshold of ≤8 g/dL is recommended for participants undergoing orthopedic surgery, cardiac surgery, and those with preexisting cardiovascular disease.
Time Frame: From Week 5 up to approximately 24 months
Population: Data were not collected for this outcome measure nor conducted as part of the final analysis as they were not deemed critical for the aCSR.
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Participants With Occurrence of Erythropoiesis-Stimulating Agent (ESA) Administration
Description: If participants experienced chemotherapy-induced anemia (hemoglobin level <10 g/dL) after receiving the first dose of study treatment, ESAs may be used per ASCO guidelines to improve hematopoietic response and reduce the likelihood of RBC transfusion.
Time Frame: Up to approximately 24 months
Population: as for outcome 10
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With Occurrence of Grade 3 and 4 Decrease of Platelets
Description: Grade 3 shows signs of mucosal bleeding, such as blood crusting in nostrils or nosebleeds, petechiae or purpura in the mouth, blood in the urine or stool, and heavy periods. Grade 4 shows signs of more severe mucosal bleeding or suspected internal bleeding, such as in the brain or lungs that requires immediate medical attention.
Time Frame: Up to approximately 24 months
Population: as for outcome 10
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Platelet Transfusions
Description: Platelet transfusion is recommended at a threshold of ≤10 x 10^9/L. Platelets should also be transfused in any participant who was bleeding with a platelet count <50 x 10^9/L (100 x 10^9/L for central nervous system or ocular bleeding).
Time Frame: Up to approximately 24 months
Population: as for outcome 10
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With Occurrence of Serious Infections
Description: Participants experienced chemotherapy-induced myelosuppression faced severe clinical consequences such as serious infections are reported.
Time Frame: Up to approximately 24 months
Population: as for outcome 10
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants Administered IV Antibiotics
Time Frame: Up to approximately 24 months
Population: as for outcome 10
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 0

16. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs) and Non-serious Adverse Events (NSAEs)
Description: AEs are defined as those events occurring or worsening after treatment has begun in the study. An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: From first administration of study treatment (Day 1) up to approximately 24 months
Population: Safety Population; included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: Count of participants
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
Number analyzed (Participants) | 30
Count of participants
  Number of Participants with Any AE | 29
  Number of Participants with Any Serious AE | 6

ADVERSE EVENTS:
Time Frame: From the first administration of study treatment (Day 1) up to the end of the study visit, approximately 132 weeks.
Description: The safety population included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Trilaciclib + Sacituzumab Govitecan-hziy
All-Cause Mortality (participants affected / at risk) | 21/30
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trilaciclib + Sacituzumab Govitecan-hziy (N=30)
Breast cellulitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Dizziness (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trilaciclib + Sacituzumab Govitecan-hziy (N=30)
Nausea (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 19
Pyrexia (General disorders) | 4
Asthenia (General disorders) | 3
Chills (General disorders) | 2
Localised oedema (General disorders) | 2
Oedema peripheral (General disorders) | 2
Headache (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 7
Dysgeusia (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 2
Restless legs syndrome (Nervous system disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Chest wall necrosis (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 11
Dry skin (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
COVID-19 (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Neutrophil count decreased (Investigations) | 7
White blood cell count decreased (Investigations) | 7
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Insomnia (Psychiatric disorders) | 7
Palpitations (Cardiac disorders) | 4
Atrial fibrillation (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 6
Anaemia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 3
Flushing (Vascular disorders) | 4
Hot flush (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Breast pain (Reproductive system and breast disorders) | 4
Fall (Injury, poisoning and procedural complications) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees to submit any disclosure to Sponsor for review at least thirty (30) days prior to submission. Within sixty (60) days of its receipt, Sponsor can provide feedback on any disclosure Sponsor may require Investigator to remove, Confidential Information (other than study data), and/or to delay the proposed publication or presentation for an additional sixty (60) days to enable Sponsor to seek patent protection for inventions.

DOCUMENTS (2):
  • Study Protocol (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT05113966/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT05113966/SAP_001.pdf